CLINICAL TRIAL: NCT05420480
Title: Two-field Versus Three-field Lymph Node Dissection for Esophageal Squamous Cell Carcinoma Patients Without Cervical Lymph Node Metastasis After Neoadjuvant Therapy: A Multi-center, Prospective Randomized Controlled Study
Brief Title: Two-field Versus Three-field Lymph Node Dissection in ESCC After Neoadjuvant Therapy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Baoji Central Hospital (Other); Sixth Affiliated Hospital, Sun Yat-sen University (Other); Suining Central Hospital (Other); Jieyang People's Hospital (Other); Second Affiliated Hospital of Nantong University (Other); Taixing People's Hospital (Other); Hebei Medical University Fourth Hospital (Other); Suzhou Municipal Hospital (Other); Fujian Provincial Hospital (Other); Jining First People's Hospital (Other); The General Hospital of Western Theater Command (Other); Zhejiang Cancer Hospital (Other); Shanghai Chest Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2022-154
Record Dates: First submitted 2022-06-12; First posted 2022-06-15 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: Esophageal Squamous Cell Carcinoma; Esophagectomy; Neoadjuvant therapy
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Two-Field lymph node dissection (106recR negative by intra-operative frozen section pathology) (Active Comparator): The right recurrent laryngeal nerve lymph node (106recR) will be dissected and subjected to the intra-operative frozen section pathology. If the 106recR lymph node has no metastasis, esophagectomy and "Two-Field" lymph node dissection will be performed.
  Interventions: Procedure: Two-Field lymph node dissection
- Three-Field lymph node dissection (106recR negative by intra-operative frozen section pathology) (Experimental): The right recurrent laryngeal nerve lymph node (106recR) will be dissected and subjected to the intra-operative frozen section pathology. If the 106recR lymph node has no metastasis, esophagectomy and "Three-Field" lymph node dissection will be performed.
  Interventions: Procedure: Three-Field lymph node dissection
- Three-Field lymph node dissection (106recR positive by intra-operative frozen section pathology) (Other): The right recurrent laryngeal nerve lymph node (106recR) will be dissected and subjected to the intra-operative frozen section pathology. If the 106recR lymph node has metastasis, esophagectomy and "Three-Field" lymph node dissection will be performed.
  Interventions: Procedure: Three-Field lymph node dissection

INTERVENTIONS:
Procedure: Two-Field lymph node dissection — The right recurrent laryngeal nerve lymph node (106recR) will be dissected and subjected to the intra-operative frozen section pathology. If the 106recR lymph node has no metastasis, patients will be randomized to two groups at 1:1 ratio and receive esophagectomy with "Two-Field" or "Three-Field" lymph node dissection.
  Arms: Two-Field lymph node dissection (106recR negative by intra-operative frozen section pathology)
Procedure: Three-Field lymph node dissection — The right recurrent laryngeal nerve lymph node (106recR) will be dissected and subjected to the intra-operative frozen section pathology. If the 106recR lymph node has no metastasis, patients will be randomized to two groups at 1:1 ratio and receive esophagectomy with "Two-Field" or "Three-Field" lymph node dissection.
  Arms: Three-Field lymph node dissection (106recR negative by intra-operative frozen section pathology)
Procedure: Three-Field lymph node dissection — The right recurrent laryngeal nerve lymph node (106recR) will be dissected and subjected to the intra-operative frozen section pathology. If the 106recR lymph node has metastasis, esophagectomy and "Three-Field" lymph node dissection will be performed.
  Arms: Three-Field lymph node dissection (106recR positive by intra-operative frozen section pathology)

SUMMARY:
Comparison of esophagectomy with Two-field Versus Three-field lymphadenectomy in locally advanced ESCC patients after neoadjuvant therapy

DETAILED DESCRIPTION:
In locally advanced esophageal squamous cell carcinoma patients, neoadjuvant therapy has become a standard therapeutic strategy and been widely administered. Neoadjuvant therapy drastically reduces the metastatic lymph nodes rate as verified in numerous studies including CROSS (Netherlands), JCOG9907/1109 (Japan), NEOCRTEC5010 and CMISG1701 (China) trials, which entails a study to characterize the distribution of lymph node metastasis, and to identify the optimal extent of lymphadenectomy in ESCC patients who received neoadjuvant therapy.

This study aims to clarify whether three-field (cervical-thoracic-abdominal) lymphadenectomy will improve survival over two-field (thoracic-abdominal) lymphadenectomy for ESCC patients after neoadjuvant therapy.

An estimated 323 patients will be enrolled. Eligible patients will undergo right recurrent laryngeal nerve lymph node dissection (106recR), which will be subjected to intra-operative frozen resection pathological evaluation. If 106recR lymph node reports POSITIVE, patients will undergo esophagectomy with Three-Field lymphadenectomy (n=75). If 106recR lymph node reports NEGATIVE, patients will be randomized at 1:1 ratio into two groups: A) Esophagectomy with Two-Field lymphadenectomy (n=124) or B) Esophagectomy with Three-Field lymphadenectomy (n=124). Analyses will be done according to the intention-to-treat principle.

The primary end point is overall survival (OS), calculated from the date of randomization to the date of death from any cause. Secondary end point is Disease-free survival. Other exploratory end points include tumor recurrence pattern, quality of life, peri-operative complications, and the correlation between metastases of 106recR and cervical lymph nodes.

ELIGIBILITY:
Inclusion Criteria:

1. Squamous cell carcinoma was diagnosed by the pathological type of gastroscopic biopsy;
2. The primary tumor is located in the thoracic, and the primary site of esophageal cancer is determined by the location of the esophagus where the upper edge of the mass is located (upper thoracic esophagus: from the entrance of the thoracic cavity, down to the level of the lower edge of the azygos vein arch, 20 cm from the incisors to the endoscopy <25 cm; middle thoracic esophagus: from the lower border of the azygos vein arch, down to the level of the inferior pulmonary vein, 25 cm to 30 cm from the incisors on endoscopy; lower thoracic esophagus: from the level of the inferior pulmonary veins, down to the stomach, internal Endoscopy 30 cm to 40 cm from the incisors);
3. According to the above examinations, patients with cII-III stage esophageal squamous cell carcinoma after received neoadjuvant therapy (including neoadjuvant chemoradiotherapy, neoadjuvant chemotherapy, neoadjuvant immunotherapy or neoadjuvant immunotherapy combined with chemotherapy, etc.), preoperative clinical evaluation was performed. Patients with esophageal cancer of clinical stage ycT1b-3N0-1M0 who can undergo surgical resection (enhanced chest and abdomen CT, cervical lymph node ultrasound and other methods to evaluate whether the tumor has obvious external invasion, whether the mediastinal lymph nodes have obvious enlargement, whether there are distant organs metastases or not); if the primary tumor is suspected to be T4b, multiple mediastinal lymph node metastases, or remote metastases, etc., whole-body PET-CT, endoscopic ultrasonography (EUS) (optional) and other tests are performed to further clarify the clinical stage), and there is no large cervical lymph nodes (<0.8 cm in short-axis diameter of lymph nodes by CT or ultrasonography, or <0.65 in short- and long-axis diameters of lymph nodes)
4. Age ≥18 years old, ≤75 years old, physical condition score ECOG 0～1, expected survival period ≥12 months;
5. No major organ dysfunction, blood routine, lung, liver, kidney and heart functions were basically normal.

   Laboratory test indicators must meet the following requirements:

   Blood: white blood cells>4.0×109/L, absolute count of neutrophils (ANC)≥2.0×109/L, platelet count>100×109/L, hemoglobin>90g/L Pulmonary function: FEV1≥1.2L, FEV1%≥50%, and DLCO≥50%; usually in elderly patients (over 60 years old), lung function is assessed by the stair climbing test; Liver function: serum bilirubin less than 1.5 times the maximum normal value; ALT and AST less than 1.5 times the maximum normal value.

   Renal function: Serum creatinine (SCr)≤120µmol/L, creatinine clearance rate (CCr)≥60ml/min;
6. Be able to understand the situation of this research and sign the informed consent.
7. No gender selection
8. No healthy subjects are accepted

Exclusion Criteria:

1. Enhanced CT of chest and abdomen, ultrasound of cervical lymph nodes, whole body PET-CT (optional) or EBUS (optional), etc.

   The clinical staging was determined by imaging examination as (AJCC/UICC8th Edition) T4b unresectable (can be treated by two judged by a senior thoracic surgeon) [52], multiple lymphadenopathy (estimated lymph node metastasis ≥ 3), multiple sites Patients with enlarged lymph nodes (estimated number of lymph node metastases ≥ 2) or distant metastasis (M1); patients with enlarged lymph nodes Cervical lymph nodes (the short-axis diameter of lymph nodes determined by CT or ultrasonography is > 0.8 cm, or the short and long diameters of lymph nodes are > 0.8 cm.

   0.65);
2. Those who have received or are receiving other chemotherapy, radiotherapy or targeted therapy;
3. The pathology of gastroscopy is non-squamous cell carcinoma;
4. Have other tumors in the past (except for those who have suffered from cervical carcinoma in situ or local skin basal cell carcinoma and have been cured); Other exclusion criteria.
5. History of autoimmune diseases;
6. recent or current use of hormones or immunosuppressants;
7. Received immunotherapy in the past;
8. Have a history of severe hypersensitivity to antibody drugs in the past;
9. Past or ongoing chronic or recurrent autoimmune disease;
10. Interstitial lung disease, pulmonary fibrosis, diverticulitis or systemic ulcerative gastrointestinal inflammation;
11. Confirmed history of congestive heart failure; angina pectoris poorly controlled by drug therapy; electrocardiogram (ECG) confirmed of transmural myocardial infarction; uncontrolled hypertension; clinically significant valvular heart disease; or high-risk uncontrolled arrhythmia;
12. Severe uncontrolled systemic interstitial diseases, such as active infection or poorly controlled diabetes; abnormal coagulation function, bleeding tendency, or receiving thrombolytic or anticoagulant therapy;
13. Women with positive serum pregnancy test or breastfeeding, and men and women of childbearing age who are unwilling to use adequate contraception during study drug treatment;
14. Known immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV) activity Sexual infection or known HIV seropositivity; including HBV or HCV surface antigen positivity (RNA);
15. Known allergy to any study drug;
16. Have a history of organ transplantation (including bone marrow autologous transplantation and peripheral stem cell transplantation);
17. Those who have peripheral nervous system disorders or a history of obvious mental disorders and central nervous system disorders;
18. Concomitant use of anti-tumor drugs outside the research protocol;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 323 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival(OS) | Up to the date of death of any causes since the date of surgery, up to 36 months

SECONDARY OUTCOMES:
Disease free survival (DFS) | Up to the date of death of any causes since the date of surgery, up to 36 months
  Disease recurrence is defined as locoregional (esophageal bed or anastomotic or regional lymph nodes) or metastatic (supraclavicular lymph nodes or distant organs)

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Zhongshan Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Torre LA, Bray F, Siegel RL, Ferlay J, Lortet-Tieulent J, Jemal A. Global cancer statistics, 2012. CA Cancer J Clin. 2015 Mar;65(2):87-108. doi: 10.3322/caac.21262. Epub 2015 Feb 4. PMID 25651787
- [Background] Chen W, Zheng R, Baade PD, Zhang S, Zeng H, Bray F, Jemal A, Yu XQ, He J. Cancer statistics in China, 2015. CA Cancer J Clin. 2016 Mar-Apr;66(2):115-32. doi: 10.3322/caac.21338. Epub 2016 Jan 25. PMID 26808342